CLINICAL TRIAL: NCT00906178
Title: CyberSenga: Harnessing the Power of the Internet to Prevent HIV in Ugandan Youth
Brief Title: CyberSenga: Internet-based HIV Prevention in Uganda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Mbarara University of Science and Technology (Other); Harvard University (Other); University of Colorado, Denver (Other); Internet Solutions for Kids Uganda, Limited (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ISK-NIH-MH080662; 5R01MH080662 (NIH)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Sexual Abstinence; Condom Use
Keywords: HIV prevention; technology; adolescent; developing countries
MeSH Terms: conditions — Sexual Abstinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CyberSenga (Experimental): 6-module HIV prevention program tailored for adolescents in Uganda
  Interventions: Behavioral: CyberSenga
- Control (No Intervention): "treatment as usual" - the sexual health education adolescents currently receive in secondary school

INTERVENTIONS:
Behavioral: CyberSenga — Internet-based HIV prevention program
  Arms: CyberSenga

SUMMARY:
The investigators propose to design and test an Internet-based HIV prevention program for adolescents in Uganda.

DETAILED DESCRIPTION:
HIV/AIDS is a major contributor to morbidity and mortality in Uganda. Despite aggressive advances in HIV prevention efforts, recent data suggest that HIV prevalence is increasing generally, and HIV knowledge, a direct contributor to behavior, is on the decline among young people specifically as compared to a decade ago.

The Internet is a promising mode of intervention delivery in resource poor-settings because the costs associated with scaling up are minimal; dissemination online is the same if one person or 100,000 people use the program. Just as important, it provides access to important health information in a stigma-free, anonymous atmosphere. Our recent data indicate that 45% of adolescents in Mbarara, Uganda have used the Internet, 78% of whom went online at least once in the previous week. Eighty-one percent of respondents in the same survey indicated they would go to an HIV prevention web site if it existed. Based upon these data, we propose to develop a culturally appropriate, Internet-based HIV prevention program designed specifically for Ugandan adolescents between the ages of 12 and 18 years. Our specific aims are as follows:

Specific Aim 1: Design a 6-hour, Internet-based HIV prevention program for adolescents. Content will be culturally tailored to the HIV preventive information, motivation, and behavioral skills needs of Ugandan adolescents.

Specific Aim 2: Test the intervention in a randomized controlled trial (n=500) among adolescents attending grades Secondary 1-4 (similar to US high school grades 8th - 11th) at day schools in Mbarara.

This project has the potential to develop low-cost and salable interventions to HIV transmission risk behaviors among adolescents in Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in grades Secondary 1 through 4 at a partner secondary school
* Having used a computer or the Internet at least once in the past year
* Not having been part of the intervention development activities
* Caregiver informed permission and adolescent informed assent

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ybarra, MPH PhD, Principal Investigator — Center for Innovative Public Health
Locations (1):
- Internet Solutions for Kids Uganda, Limited, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell KJ, Bull S, Kiwanuka J, Ybarra ML. Cell phone usage among adolescents in Uganda: acceptability for relaying health information. Health Educ Res. 2011 Oct;26(5):770-81. doi: 10.1093/her/cyr022. Epub 2011 May 2. PMID 21536715
- [Background] Bull S, Nabembezi D, Birungi R, Kiwanuka J, Ybarra M. Cyber-Senga: Ugandan youth preferences for content in an internet-delivered comprehensive sexuality education programme. East Afr J Public Health. 2010 Mar;7(1):58-63. PMID 21413574
- [Background] Ybarra ML, Biringi R, Prescott T, Bull SS. Usability and navigability of an HIV/AIDS internet intervention for adolescents in a resource-limited setting. Comput Inform Nurs. 2012 Nov;30(11):587-95; quiz 596-7. doi: 10.1097/NXN.0b013e318266cb0e. PMID 22918136
- [Background] Hampanda K, Ybarra M, Bull S. Perceptions of health care services and HIV-related health-seeking behavior among Uganda adolescents. AIDS Care. 2014;26(10):1209-17. doi: 10.1080/09540121.2014.894612. Epub 2014 Mar 13. PMID 24625122
- [Background] Ybarra ML, Korchmaros J, Kiwanuka J, Bangsberg DR, Bull S. Examining the applicability of the IMB model in predicting condom use among sexually active secondary school students in Mbarara, Uganda. AIDS Behav. 2013 Mar;17(3):1116-28. doi: 10.1007/s10461-012-0137-x. PMID 22350827
- [Background] Katz IT, Ybarra ML, Wyatt MA, Kiwanuka JP, Bangsberg DR, Ware NC. Socio-cultural and economic antecedents of adolescent sexual decision-making and HIV-risk in rural Uganda. AIDS Care. 2013;25(2):258-64. doi: 10.1080/09540121.2012.701718. Epub 2012 Jul 27. PMID 22835224
- [Background] Ybarra ML, Bull SS, Kiwanuka J, Bangsberg DR, Korchmaros J. Prevalence rates of sexual coercion victimization and perpetration among Uganda adolescents. AIDS Care. 2012;24(11):1392-400. doi: 10.1080/09540121.2011.648604. Epub 2012 Feb 2. PMID 22299764
- [Background] Birungi R, Nabembezi D, Kiwanuka J, Ybarra M, Bull S. Adolescents' perceptions of sexual coercion in Uganda. Afr J AIDS Res. 2011 Dec;10(4):487-94. doi: 10.2989/16085906.2011.646664. PMID 25865380
- [Background] Ybarra ML, Emenyonu N, Nansera D, Kiwanuka J, Bangsberg DR. Health information seeking among Mbararan adolescents: results from the Uganda Media and You survey. Health Educ Res. 2008 Apr;23(2):249-58. doi: 10.1093/her/cym026. Epub 2007 Jul 16. PMID 17639121
- [Result] Ybarra ML, Korchmaros JD, Prescott TL, Birungi R. A Randomized Controlled Trial to Increase HIV Preventive Information, Motivation, and Behavioral Skills in Ugandan Adolescents. Ann Behav Med. 2015 Jun;49(3):473-85. doi: 10.1007/s12160-014-9673-0. PMID 25633626
- [Result] Ybarra ML, Bull SS, Prescott TL, Birungi R. Acceptability and feasibility of CyberSenga: an Internet-based HIV-prevention program for adolescents in Mbarara, Uganda. AIDS Care. 2014 Apr;26(4):441-7. doi: 10.1080/09540121.2013.841837. Epub 2013 Oct 4. PMID 24093828
- [Result] Ybarra ML, Bull SS, Prescott TL, Korchmaros JD, Bangsberg DR, Kiwanuka JP. Adolescent abstinence and unprotected sex in CyberSenga, an Internet-based HIV prevention program: randomized clinical trial of efficacy. PLoS One. 2013 Aug 14;8(8):e70083. doi: 10.1371/journal.pone.0070083. eCollection 2013. PMID 23967069
- Available data/document: Intervention website — http://www.cybersenga.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We aimed to screen all 382 female students enrolled in the two mixed-sex schools and 772 of the 2,264 male students enrolled across the four schools to identify 400 eligible youth. Many youth were out of school trying to secure school fees or had changed schools. As a result, 740 of the youth were screened, 416 of whom were eligible (56%).
Groups:
- HIV Prevention: 6-module HIV prevention program tailored for adolescents in Uganda
  CybereSenga: Internet-based HIV prevention program
- Control: "treatment as usual" - the sexual health education adolescents currently receive in secondary school
  CybereSenga: Internet-based HIV prevention program
Period: Overall Study
Arm/Group | HIV Prevention | Control
Started | 183 | 183
Completed | 168 | 167
Not Completed | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Prevention | Control | Total
Number analyzed (Participants) | 183 | 183 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.4) | 16.2 (1.5) | 16.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 152 | 155 | 307
Grade [Number; unit: participants]
  Secondary 2 | 47 | 50 | 97
  Secondary 3 | 73 | 58 | 131
  Secondary 4 | 63 | 75 | 138
Maternal Education [Number; unit: participants]
  Primary School or Less/Don't Know | 60 | 63 | 123
  More Than Primary School | 123 | 120 | 243
Paternal Education [Number; unit: participants]
  Primary School or Less/Don't Know | 48 | 50 | 98
  More Than Primary School | 135 | 133 | 268
Internet Use [Number; unit: participants]
  Infrequent | 101 | 102 | 203
  Frequent | 82 | 81 | 163
Ever Had Oral Sex [Number; unit: participants]
  Yes | 19 | 17 | 36
  No | 164 | 166 | 330
Ever Had Vaginal Sex [Number; unit: participants]
  Yes | 58 | 55 | 113
  No | 125 | 128 | 253
Ever Had Anal Sex [Number; unit: participants]
  Yes | 4 | 5 | 9
  No | 179 | 178 | 357
Ever Been Tested for HIV [Number; unit: participants]
  Yes | 75 | 64 | 139
  No | 108 | 119 | 227
Ever known someone who died from AIDS [Number; unit: participants]
  Yes | 67 | 71 | 138
  No | 116 | 112 | 228
Tired of hearing about HIV prevention information [Number; unit: participants]
  Somewhat/strongly agree | 45 | 49 | 94
  Do not Somewhat/strongly agree | 138 | 134 | 272
Above average change of getting HIV [Number; unit: participants] — Self-appraisal of one's likelihood of getting HIV
  participants
    Yes | 12 | 12 | 24
    No | 171 | 171 | 342
Beliefs supportive of HIV Stigma [Mean (Standard Deviation); unit: units on a scale] — This measure has a range from 0 to 4 with higher scores reflecting greater HIV stigma
  units on a scale | 1.1 (.9) | 1.2 (1.1) | 1.1 (1.0)
Ever had a boyfriend/girlfriend [Number; unit: participants]
  Yes | 141 | 137 | 278
  No | 42 | 46 | 88
Ever been a victim of teen dating violence [Number; unit: participants]
  Yes | 35 | 43 | 78
  No | 148 | 140 | 288
Ever been a perpetrator of teen dating violence [Number; unit: participants]
  Yes | 28 | 37 | 65
  No | 155 | 146 | 301
Beliefs consistent with female empowerment in relationships [Mean (Standard Deviation); unit: units on a scale] — This measure has scores that can range from 2 to 10 with higher scores being higher in these beliefs
  units on a scale | 8.2 (2.8) | 8.0 (2.8) | 8.1 (2.8)
Fair or poor health [Number; unit: participants]
  Yes | 35 | 24 | 59
  No | 148 | 159 | 307
Bright future somewhat/very unlikely [Number; unit: participants] — subject chose between somewhat likely and very likely
  participants
    Yes | 20 | 15 | 35
    No | 163 | 168 | 331
Wish to have more self-respect [Number; unit: participants]
  Yes | 149 | 144 | 293
  No | 34 | 39 | 73
The Multidimensional Scale of Perceived Social Support : Social support from "special person" [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 20 with higher scores reflecting more support
  units on a scale | 16.7 (2.8) | 16.2 (4.1) | 16.5 (4.0)
The Multidimensional Scale of Perceived Social Support: Social support from family [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 20 with higher scores reflecting more support
  units on a scale | 17.1 (3.1) | 17.7 (3.0) | 17.4 (3.1)
Information [Number; unit: participants] — 80% or more answers about HIV correct
  participants
    Yes | 86 | 97 | 183
    No | 97 | 86 | 183
Motivation: Attitudes towards HIV preventive acts [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 5 with higher scores reflecting more motivation
  units on a scale | 3.6 (.9) | 3.5 (.9) | 3.6 (.9)
Motivation: Subjective norms regarding HIV preventive acts [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 5 with higher scores reflecting more motivation
  units on a scale | 3.6 (.9) | 3.5 (.9) | 3.6 (.9)
Motivation: Behavioral intentions for HIV prevention [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 5 with higher scores reflecting more motivation
  units on a scale | 3.5 (.9) | 3.5 (.9) | 3.5 (.9)
Behavioral Skills [Mean (Standard Deviation); unit: units on a scale] — This measure has scores possibly ranging form 1 to 5 with higher scores reflecting more skills
  units on a scale | 2.9 (.7) | 2.9 (.7) | 2.9 (.7)

OUTCOME MEASURES:

1. Primary Outcome: Sex Without a Condom as Assessed by Self-report
Description: Unprotected sex (i.e., vaginal or anal sex without a condom) in the past three months
Time Frame: 6-months post-intervention
Population: ITT - Intention to Treat
Measure: Number; unit: participants
Arm/Group | HIV Prevention | Control
Number analyzed (Participants) | 183 | 183
participants | 26 | 24
Statistical Analysis 1: Comparison: HIV Prevention vs Control; Test type: Superiority or Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [.57 to 1.94]

2. Primary Outcome: Sexual Abstinence
Description: Not having had vaginal or anal sex in the past three months
Time Frame: 6-months post-intervention
Population: ITT - Intention to Treat
Measure: Number; unit: participants
Arm/Group | HIV Prevention | Control
Number analyzed (Participants) | 183 | 183
participants | 138 | 137
Statistical Analysis 1: Comparison: HIV Prevention vs Control; Test type: Superiority or Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [.62 to 1.65]

3. Secondary Outcome: Abstinence at Three-month Follow-up
Description: Sexual abstinence (i.e., not having vaginal or anal sex) in the past 90 days
Time Frame: 3 months post-intervention
Population: ITT--Intention to Treat
Measure: Number; unit: participants
Arm/Group | HIV Prevention | Control
Number analyzed (Participants) | 183 | 183
participants | 135 | 149
Statistical Analysis 1: Comparison: HIV Prevention vs Control; Test type: Superiority or Other; Odds Ratio (OR) = 1.56, 95% CI 2-sided [.93 to 2.62]

4. Secondary Outcome: Unprotected Sex at Three-month Follow-up
Description: Ever had vaginal or anal sex without a condom in the past 90 days
Time Frame: 3 months post-intervention
Population: ITT--Intention to Treat
Measure: Number; unit: participants
Arm/Group | HIV Prevention | Control
Number analyzed (Participants) | 183 | 183
participants | 21 | 28
Statistical Analysis 1: Comparison: HIV Prevention vs Control; Test type: Superiority or Other; Odds Ratio (OR) = .70, 95% CI 2-sided [.37 to 1.30]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the study period (i.e., from baseline to 6 month follow-up).
Arm/Group | HIV Prevention | Control
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/183
Other Adverse Events (participants affected / at risk) | 0/183 | 0/183

LIMITATIONS AND CAVEATS:
Sexual activity in adolescence is a stigmatized behavior in Uganda, especially for females. Youth may have under-reported their sexual experiences, which in the intervention group would have led to them being triaged to the incorrect content.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No